CLINICAL TRIAL: NCT02642874
Title: Methocarbamol in Treatment of Muscle Cramps in Cirrhotic Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Consultant liver and GIT diseases- Tanta university hospital, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: methocarbamol
Record Dates: First submitted 2015-12-25; First posted 2015-12-30 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Methocarbamol; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methocarbamol (Experimental): Methocarbamol twice daily
  Interventions: Drug: Methocarbamol
- placebo (Placebo Comparator): Calcium carbonate twice daily
  Interventions: Drug: Calcium Carbonate

INTERVENTIONS:
Drug: Methocarbamol — Methocarbamol twice daily
  Other Names: Flexpro
  Arms: Methocarbamol
Drug: Calcium Carbonate — Calcium carbonate twice daily
  Other Names: Calcitron
  Arms: placebo

SUMMARY:
Muscle cramps markedly affect the quality of life in cirrhotic patients with no highly effective drug. Methocarbamol is a central muscle relaxant used to treat skeletal muscle spasms. The mechanism of action of methocarbamol is currently unknown, but may involve the inhibition of carbonic anhydrase. Methocarbamol has a high therapeutic index, i.e. a wide range of safe and effective dosages.

DETAILED DESCRIPTION:
Muscle cramps markedly affect the quality of life in cirrhotic patients with no highly effective drug. Abrams et al compared patients with cirrhosis with those with congestive heart failure and found a significantly higher prevalence of weekly or daily cramps with cirrhosis (22%) vs patients with congestive heart failure (5%). Interestingly, there was no difference in diuretic use or dosing between the 2 groups, supporting that factors other than diuretic-mediated effects explained the differences. Methocarbamol is a central muscle relaxant used to treat skeletal muscle spasms. The mechanism of action of methocarbamol is currently unknown, but may involve the inhibition of carbonic anhydrase. Methocarbamol has a high therapeutic index, i.e. a wide range of safe and effective dosages.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients with frequent muscle cramps.

Exclusion Criteria:

* Elderly patients.
* Encephalopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
number of muscle cramps | 3 months
  change in number of muscle cramps

CONTACTS AND LOCATIONS:
Overall Officials: Sherief M. Abd-Elsalam, Consultant, Principal Investigator — liver diseases dept.- Tanta university hospital; Walaa A. Elkhalawany, Consultant, Study Director — liver diseases dept.- Tanta university hospital
Locations (1):
- Tanta university - faculty of medicine, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided